CLINICAL TRIAL: NCT01014221
Title: Acupuncture in Patients With Carpal Tunnel Syndrome ~ A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuang Tien General Hospital (Other)
Responsible Party: Yang, chun-pai/ Attending physician of Department of Neurology, Kuang Tien General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9612
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Carpal Tunnel Syndrome
Keywords: acupuncture; carpal tunnel syndrome; CTS; steroid; global symptom score (GSS)
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Acupuncture Therapy; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture group (Experimental): acupuncture administered in 8 sessions over 4 weeks
  Interventions: Other: Acupuncture
- Steroid group (Active Comparator): 2 weeks of prednisolone 20 mg daily followed by 2 weeks of prednisolone 10 mg daily
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Other: Acupuncture — acupuncture administered in 8 sessions over 4 weeks
  Arms: Acupuncture group
Drug: Prednisolone — 2 weeks of prednisolone 20 mg daily followed by 2 weeks of prednisolone 10 mg daily
  Arms: Steroid group

SUMMARY:
To investigate the efficacy of acupuncture compared with steroid treatment in patients with mild-to-moderate carpal tunnel syndrome (CTS) as measured by objective changes in nerve conduction studies (NCS) and subjective symptoms assessment in a randomized, controlled study.

DETAILED DESCRIPTION:
A total of 77 consecutive and prospective CTS patients confirmed by NCS were enrolled in the study. Those who had fixed sensory complaint over the median nerve and thenar muscle atrophy were excluded. The CTS patients were randomly divided into 2 treatment arms: (1) 2 weeks of prednisolone 20 mg daily followed by 2 weeks of prednisolone 10 mg daily (n =39), and (2)acupuncture administered in 8 sessions over 4 weeks (n=38). A validated standard questionnaire as a subjective measurement was used to rate the 5 major symptoms (pain, numbness, paresthesia,weakness/clumsiness, and nocturnal awakening) on a scale from 0 (no symptoms) to 10 (very severe). The total score in each of the 5 categories was termed the global symptom score (GSS). Patients completed standard questionnaires at baseline and 2 and 4 weeks later. The changes in GSS were analyzed to evaluate the statistical significance. NCS were performed at baseline and repeated at the end of the study to assess improvement. All main analyses used intent-to-treat.

ELIGIBILITY:
Inclusion Criteria:

presence of at least one of the following primary symptoms:

1. numbness, tingling pain, or paresthesia in the median nerve distribution;
2. precipitation of these symptoms by repetitive hand activities, which could be relieved by resting, rubbing, and shaking the hand; and
3. nocturnal awakening by such sensory symptoms.- plus the presence of 1 or more of the following standard electrophysiologic criteria:

   * (1) prolonged distal motor latency (DML) to the abductor pollicis brevis (APB)(abnormal Z4.7 ms, stimulation over the wrist, 8 cm proximal to the active electrode);
   * (2) prolonged antidromic distal sensory latency (DSL) to the second digit (abnormal Z3.1 ms; stimulation over the wrist, 14 cm proximal to the active electrode); and
   * (3) prolonged antidromic wrist-palm sensory nerve conduction velocity (W-P SNCV) at a distance of 8 cm (W-P SNCV, abnormal <45 m/s).

Exclusion Criteria:

1. symptoms occurring less than 3 months before the study or symptoms improving during the 1-month initial observation period (to exclude patients who might have spontaneous resolution of symptoms);
2. severe CTS that had progressed to visible muscle atrophy;
3. in our study, mild CTS referred to patients with decreased conduction velocity over the palm-wrist segment and delayed DSL, with normal median SNAP amplitude and CMAP amplitude of the APB. Moderate CTS referred to patients with abnormally delayed DML and DSL with either decreased median SNAP amplitude or decreased CMAP amplitude of the APB muscle. Thus, CTS patients with the presence of either fibrillation potentials or reinnervation on needle EMG in the APB were excluded (to ensure the inclusion of only mildly or moderately affected individuals);
4. clinical or electrophysiologic evidence of accompanying conditions that could mimic CTS or interfere with its evaluation, such as cervical radiculopathy, proximal median neuropathy, or significant polyneuropathy;
5. evidence of obvious underlying causes of CTS such as diabetes mellitus, rheumatoid arthritis, hypothyroidism (acromegaly), pregnancy, alcohol abuse or drug usage (steroids or drugs acting through the central nervous system), use of vibrating machinery, and suspected malignancy or inflammation or autoimmune disease were documented as underlying causes for CTS;
6. recent peptic ulcer or history of steroid intolerance;
7. prior unpleasant experience with acupuncture or a bleeding diathesis; or
8. cognitive impairment interfering with the patient's ability to follow instructions and describe symptoms.-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Global symptoms score (GSS) | Baseline, Month 1, 7, and 13

SECONDARY OUTCOMES:
eletrophysiological parameters | baseline, month 1 and 13

CONTACTS AND LOCATIONS:
Locations (1):
- Kuang Tien General Hospital, Taichung County, Taiwan, Taiwan

REFERENCES:
- [Result] Yang CP, Hsieh CL, Wang NH, Li TC, Hwang KL, Yu SC, Chang MH. Acupuncture in patients with carpal tunnel syndrome: A randomized controlled trial. Clin J Pain. 2009 May;25(4):327-33. doi: 10.1097/AJP.0b013e318190511c. PMID 19590482
- [Derived] Yang CP, Wang NH, Li TC, Hsieh CL, Chang HH, Hwang KL, Ko WS, Chang MH. A randomized clinical trial of acupuncture versus oral steroids for carpal tunnel syndrome: a long-term follow-up. J Pain. 2011 Feb;12(2):272-9. doi: 10.1016/j.jpain.2010.09.001. Epub 2010 Nov 26. PMID 21111685